CLINICAL TRIAL: NCT06601621
Title: Study on the Impact of Electroacupuncture Combined With Self-Acupressure on the Quality of Life of Patients With Early-Stage Breast Cancer Undergoing Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiuda Zhao (Other)
Responsible Party: Sponsor-Investigator, Jiuda Zhao, Breast Disease Diagnosis and Treatment Center, Affiliated Hospital of Qinghai University
Organization: Affiliated Hospital of Qinghai University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHQU-2024002
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Electroacupuncture; Quality of Life (QOL); Acupressure; Breast Cancer; Chemotherapy
Keywords: electroacupuncture; self-acupressure; Quality of life (QOL); breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True electroacupuncture + True self-acupressure (Experimental): Participants will receive two electroacupuncture treatments during the first week of the chemotherapy cycle. The acupuncturist will insert needles into the acupoints and manipulate the needles until"de qi"sensation is achieved and reported by the participants. Electrical stimulation will be delivered for 30 minutes at alternating frequencies of 2/10Hz. Participants will do acupressure daily during the second week of the chemotherapy cycle (two weeks for one chemotherapy cycle) or the second and third weeks (three weeks for one chemotherapy cycle). participants performed true self-acupressure, pressing each acupoint with their thumb to achieve "deqi" for three minutes.
  Interventions: Combination Product: electroacupuncture+ self-acupressure
- Sham electroacupuncture + Sham self-acupressure (Placebo Comparator): The sham acupuncture is the use of minimally invasive shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive minimal acupuncture treatment without electrical stimulation at the same time as the intervention group. Care was taken to avoid "de qi" sensation. Sham self-acupressure: Administered non-acupressure points 1 to 3cm away from the true acupressure points used in the experimental group and away from known meridians. The frequency, course duration, and overall treatment time will be the same as those in the true self-administered shiatsu group. The applied pressure does not cause a feeling of "deqi".
  Interventions: Combination Product: sham electroacupuncture + sham self-acupressure

INTERVENTIONS:
Combination Product: electroacupuncture+ self-acupressure — Participants will receive two electroacupuncture treatments within the first week of each treatment cycle. The acupuncturist inserts the needle into the point and manipulates the needle until the feeling of "deqi"; is achieved and reported by the participant. The electrical stimulation will be administered at a sustained frequency of 2/10Hz for 30 minutes. self-acupressure: In weeks 2 and 3 of each treatment cycle, participants performed true self-administered acupressure, pressing each acupoint with their thumb to achieve "deqi"; for three minutes.
  Arms: True electroacupuncture + True self-acupressure
Combination Product: sham electroacupuncture + sham self-acupressure — Sham electroacupuncture: The sham electroacupuncture shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive acupuncture treatment without electrical stimulation same the intervention group. And avoid "deqi"; sensation. Sham self-acupressure: Administered non-acupressure points 1 to 3cm away from the true acupressure points used in the experimental group and away from known meridians. The frequency, course duration, and overall treatment time will be the same as those in the true self-administered shiatsu group. The applied pressure does not cause a feeling of "deqi".
  Arms: Sham electroacupuncture + Sham self-acupressure

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effect of electroacupuncture combined with self-acupressure on the quality of life of early-stage breast cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
This study is a parallel-group, blinded (participant, evaluator, and statisticians), randomized controlled trial to investigate the effect of electroacupuncture combined with self-acupressure on the quality of life of early-stage breast cancer patients receiving chemotherapy. Patients in each group will receive electroacupuncture or sham electroacupuncture during the first week of the chemotherapy cycle. They will receive self-acupressure or sham acupressure during the second and third weeks of the chemotherapy cycle. Participants will be asked to complete the EQ-5D-5L and FACT-B scales. Primary and secondary outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and aged 75 years or younger, inclusive. with an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
2. Patients who have not received prior chemotherapy and are scheduled to receive at least 4 cycles of adjuvant or neoadjuvant chemotherapy or combination targeted therapy;
3. Normal organ function with platelets ≥ 100*10^9/ L, hemoglobin ≥ 90 g/L, serum creatinine ≤ 1.5 mg/dl (133 mmol/L), or creatinine clearance ≥ 60 ml/min, total bilirubin ≤ 1.5 times the upper limit of normal (ULN), alanine aminotransferase ≤ 2.5 times ULN, and aspartate aminotransferase ≤ 2.5 times ULN;
4. Premenopausal women need appropriate contraception;
5. Ability to understand the study well and complete the study questionnaire.

Exclusion Criteria:

1. Patients with needle phobia or allergy to stainless steel needles; and
2. Current diagnosis of mental illness (e.g., major depression, obsessive-compulsive disorder, or schizophrenia);
3. History of autoimmune diseases, blood disorders, or organ transplantation, or long-term use of hormones or immunosuppressants;
4. Comorbid bleeding disorders or thyroid dysfunction;
5. Implantation of a pacemaker; pregnancy or breastfeeding;
6. A plan for adjuvant radiotherapy in the upcoming chemotherapy cycle;
7. Current active infection;
8. Acupuncture treatment within the last four weeks;
9. Patients who are allergic to the drugs used;
10. Use of other Traditional Chinese Medicine (TCM) techniques such as Chinese herbs in the next chemotherapy cycle.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-10-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Differences in quality of life during the overall stage | Chemotherapy treatment was initiated to 21 days after the last chemotherapy cycle
  Difference in change in EQ-5D-5L scores from first to last assessment between two arms

SECONDARY OUTCOMES:
Differences in quality of life during the overall stage | Chemotherapy treatment was initiated to 21 days after the last chemotherapy cycle
  Difference in change in FACT-B scores from first to last assessment between two arms
Changes in scores on the five dimensions of the EQ-5D-5L | Chemotherapy treatment was initiated to 21 days after the last chemotherapy cycle
  Changes in mobility, self-care, daily activities, pain/discomfort,anxiety/depression before and after chemotherapy.
Changes in the dimensions of the FACT-B scale | Chemotherapy treatment was initiated to 21 days after the last chemotherapy cycle
  Physical functioning, social/family functioning, emotional functioning and functional status before and after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China